CLINICAL TRIAL: NCT04220970
Title: Breast Implant-associated Anaplastic Large Cell Lymphoma (BIA-ALCL) Registry
Status: Recruiting | Type: Observational
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Other Study IDs: BIA-ALCL Registry
Record Dates: First submitted 2020-01-06; First posted 2020-01-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Anaplastic Large Cell Lymphoma Associated With Breast Implants (BIA-ALCL)
Keywords: BIA-ALCL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 13 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BIA-ALCL
  Interventions: Other: BIA-ALCL

INTERVENTIONS:
Other: BIA-ALCL — Observational : no intervention

SUMMARY:
Anaplastic large cell lymphoma associated with breast implants (BIA-ALCL) is a rare disease seen only in women with a breast implant.

Because of the low incidence of this disease and the peculiar histological subtype, French authorities, in accordance with the recommendations of an expert group, recommended the implementation of a BIA-ALCL case registry, in connection with a national Multidisciplinary meeting (Réunion de Concertation Pluridisciplinaire nationale de recours- RCP).

This registry is opened in France and in Belgium

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with an anaplastic large cell lymphoma associated with breast implants

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female with Breast implants
Study Population: Adult patients with an anaplastic large cell lymphoma associated with breast implants
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-06-07 (Actual); Primary Completion 2032-06-07 (Estimated); Study Completion 2032-06-07 (Estimated)

PRIMARY OUTCOMES:
Overall response | 13 years

CONTACTS AND LOCATIONS:
Locations (31):
- Belgium (10):
  - A. Z. Sint-Jan Brugge-Oostende AV, Bruges
  - Clinique Universitaire Saint LUC, Brussels
  - Cliniques Universitaires de Bruxelles - Hôpital Erasme, Brussels
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
  - CHU de Liège -Domaine Sart Tilman, Liège
  - CHU UCL Namur - Site Godinne, Yvoir
- France (21):
  - CH d Avignon - Hopital Henri Duffaut, Avignon
  - Institut Bergonié, Bordeaux
  - CHRU de Brest - Hôpital Morvan, Brest
  - Hopital Louis Pasteur, Colmar
  - APHP - Hopital Henri Mondor, Créteil
  - CHU de Dijon - Hôpital le Bocage, Dijon
  - Centre Médical la Roseraie, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CH Saint-Eloi, Montpellier
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Hôpital Cochin, Paris
  - CH de Pau, Pau
  - CH de Perpigan, Perpignan
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Chu de Reims - Hopital Robert Debre, Reims
  - Centre Henri Becquerel, Rouen
  - Centre Rene Hugenin, Saint-Cloud
  - CH de Saint Malo, St-Malo
  - CHRU de Strasbourg, Strasbourg
  - Institut Universitaire du Cancer - Oncopole Toulouse (IUCT-O), Toulouse

IPD SHARING:
Plan to Share IPD: No